CLINICAL TRIAL: NCT05982405
Title: Long-term Effects of Inspiratory Muscle Training in Individuals With Chronic Venous Insufficiency
Brief Title: Long-term Effects of Inspiratory Muscle Training in Chronic Venous Insufficiency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients could not be reached for long-term follow-up.
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Assoc. prof, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Long effects of IMT
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Venous Insufficiency
Keywords: Venous Insufficiency; pain; edema; respiratory function tests; maximal respiratory pressures; exercise capacity; quality of life
MeSH Terms: conditions — Venous Insufficiency; Pain; Edema

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The individuals in the training group will be performed inspiratory muscle training using an inspiratory muscle training device (PowerBreathe®) at 30-50% of the maximal inspiratory pressure.
  Interventions: Other: Training group: Inspiratory muscle training
- Control group (Sham Comparator): Individuals in the control group will be performed thoracic expansion exercises.
  Interventions: Other: Control group: Thoracic expansion exercise

INTERVENTIONS:
Other: Training group: Inspiratory muscle training — The individuals in the training group will be performed inspiratory muscle training at 30-50% of the maximal inspiratory pressure. Inspiratory muscle training will be done using an inspiratory muscle training device (PowerBreathe®) that works with the threshold loading principle. Inspiratory muscle training will be done for 15 minutes per a session, 2 times per a day or, if tolerated, 30 minutes per a day and 1 time per a day, 5-7 days/week (one session under the supervision and the others at home), for a total of 6 weeks. Applications made at home will be followed with a diary.
  Other Names: Experimental: Training group
  Arms: Training group
Other: Control group: Thoracic expansion exercise — Individuals in the control group will be performed thoracic expansion exercises. Thoracic expansion exercises will be applied to individuals in an upright sitting position. In this position, individuals will place their hands on their lower ribs and then perform the cycle of "deep breathing + holding the deep breath for 3 seconds + slowly emptying all the breath" 3 times in a row. After this cycle, individuals will be asked to rest by taking 3-4 calm breaths. Immediately after, the individual will be asked to repeat the same cycle and repeat the cycle with calm breaths and rest until it reaches 10 repetitions. The individual will do this session 4 times a day. Individuals will do the first session of breathing exercises under supervision. In this way, incorrect exercise will be prevented. Other breathing exercise sessions will be done by individuals as a home program every day and 4 sessions a day during 6 weeks.
  Other Names: Sham Comparator: Control group
  Arms: Control group

SUMMARY:
The long-term effectiveness of inspiratory muscle training, which is known in the literature to help venous return by increasing the pump effect of the diaphragm muscle, remains unclear in individuals with chronic venous insufficiency. For this reason, in this study, it was aimed to investigate the long-term results of inspiratory muscle training in individuals with chronic venous insufficiency.

DETAILED DESCRIPTION:
Initial treatment of chronic venous insufficiency (CVI) includes conservative methods such as reducing symptoms and helping to prevent secondary problems and disease progression. If conservative methods fail, further treatments based on anatomical and physiological pathophysiological features should be applied. Treatment of CVI ranges from simple compression stockings to very complicated venous reconstructions. Physiotherapy applications also have an important place in the treatment of CVI and contain patient education, complex decongestive physiotherapy, intermittent pneumatic compression, compression garment, venous exercise programs, biomechanical stimulation therapy, proprioceptive neuromuscular facilitation, relaxation techniques and hydrotherapy methods.

Researches investigating the effectiveness of new physiotherapy applications in CVI are very limited. In one of these publications, the effects of inspiratory muscle training (IMT) and calf muscle exercise training (CMET) applied in addition to compression therapy (CT) on quality of life (QoL), venous filling time, disease severity, pain, edema, range of motion, muscle strength and functionality were investigated newly. IMT and CT were applied in group 1, CMET and CT were applied in group 2, and only CT was applied in group 3. As a result, groups of 1 and 2 showed more improvement in these outcomes compared to other groups. Acute effects of inspiratory muscle training in CVI was only shown in this study. The long-term effectiveness of inspiratory muscle training is still unclear in individuals with CVI. Therefore, this study aimed to investigate the long-term results of inspiratory muscle training in individuals with CVI.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Volunteering to participate in the study
* Diagnosed with chronic venous insufficiency using duplex ultrasound and being under standard medical treatment follow-up
* Being in one of the C1, C2, C3, C4 or C5 stages according to the Clinical, Etiology, Anatomy and Pathophysiology (CEAP) classification

Exclusion Criteria:

* Acute deep vein thrombosis, active ulcers, psychiatric disorder requiring prior vessel ablation and/or prescription drug therapy,
* Any history of chronic disease or deep vein thrombosis that may interfere with exercise capacity measurement,
* Having SARS-CoV-2 (COVID-19) or any acute infection,
* Being pregnant,
* History of arterial disease,
* Having advanced cardiorespiratory diseases, acute ulcer (< 3 months) and diabetic ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | After 6-week training and 3 months after 6-week training ends.
  The MIP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.

SECONDARY OUTCOMES:
Maximal expiratory pressure (MEP) | After 6-week training and 3 months after 6-week training ends.
  The MEP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.
Forced vital capacity (FVC) | After 6-week training and 3 months after 6-week training ends.
  Pulmonary function (Forced vital capacity (FVC)) will be evaluated with a spirometer.
Forced expiratory volume in the first second (FEV1) | After 6-week training and 3 months after 6-week training ends.
  Pulmonary function (Forced expiratory volume in the first second (FEV1)) will be evaluated with a spirometer.
FEV1 / FVC | After 6-week training and 3 months after 6-week training ends.
  Pulmonary function (FEV1 / FVC) will be evaluated with a spirometer.
Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | After 6-week training and 3 months after 6-week training ends.
  Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) will be evaluated with a spirometer.
Peak flow rate (PEF) | After 6-week training and 3 months after 6-week training ends.
  Pulmonary function (Peak flow rate (PEF)) will be evaluated with a spirometer.
Pain Intensity measured with the Numerical Rating Scale. | After 6-week training and 3 months after 6-week training ends.
  Pain intensity will be measured with the Numerical Rating Scale. This scale expresses the severity of pain with integers from 0 (no pain) to 10 (the worst possible pain).
Aerobic capacity | After 6-week training and 3 months after 6-week training ends.
  The six-minute walk test (6-MWT) will be performed according to the criteria of the American Thoracic Society for the evaluation of aerobic capacity.
Lower extremity strength | After 6-week training and 3 months after 6-week training ends.
  To determine lower extremity strength and functional mobility, the 30-second Sit-Up Test will be used in the chair.
Total quality of life score evaluated by Chronic Venous Disease Quality of Life Questionnaire | After 6-week training and 3 months after 6-week training ends.
  The score will be evaluated using Chronic Venous Disease Quality of Life Questionnaire. Each question is scored on a 5-item Likert scale. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc. Dr., Study Director — Izmir Democracy University; ÖZLEM ÇİNAR ÖZDEMİR, Assoc. Dr., Principal Investigator — Izmir Democracy University; CEMRE GÖRÜNMEZOĞLU, MSc, Principal Investigator — Izmir Democracy University; DÜNDAR ÖZALP KARABAY, Prof. Dr., Principal Investigator — Dokuz Eylul University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin G, Yeldan I, Akgul A, Ipek G. Effects of inspiratory muscle training versus calf muscle training on quality of life, pain, venous function and activity in patients with chronic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1137-1146. doi: 10.1016/j.jvsv.2022.04.012. Epub 2022 Jun 14. PMID 35710091
- [Background] Weiss RA, Munavalli G. Endovenous ablation of truncal veins. Semin Cutan Med Surg. 2005 Dec;24(4):193-9. doi: 10.1016/j.sder.2005.10.006. PMID 16387263
- [Background] Eberhardt RT, Raffetto JD. Chronic venous insufficiency. Circulation. 2005 May 10;111(18):2398-409. doi: 10.1161/01.CIR.0000164199.72440.08. No abstract available. PMID 15883226